CLINICAL TRIAL: NCT06254352
Title: Evaluation of Clinical Risk Scores in Prediction of Outcome of Acute Upper Gastrointestinal Bleeding in Non Cirrhotic Patients
Brief Title: Clinical Risk Scores in Prediction Outcome of Acute UGIT Bleeding in Non Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Abd Elaal, principal investigator, Assiut University
Other Study IDs: non variceal UGIT bleeding
Record Dates: First submitted 2024-01-15; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: scoring system — Clinical Risk Scores in Prediction of Outcome of Acute Upper Gastrointestinal Bleeding in Non Cirrhotic Patients.

SUMMARY:
To compare the ability of 4 bleeding risk scoring systems (Glasgow -Blatchford score, MAP, H3B2 and ABC scores ) in prediction of: Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay

DETAILED DESCRIPTION:
Acute upper gastrointestinal bleeding (UGIB) is a common medical emergency which has a variceal and non-variceal etiology. The non variceal etiology has higher incidence in many countries. In Egypt, non-variceal causes ranged from 26.1% to 61.6% among UGIB cases presented to the emergency departments of different University Hospitals. Guidelines recommend risk stratification early in the management of patients with acute UGIB to help triage patients into the appropriate level of care. Many scoring systems for UGIB were developed and validated from 1990s onwards. Their primary aim was to segregate the patients into low-risk and high-risk groups. High risk patients with UGIB includes those who reach some or all of the endpoints: requirement of blood transfusion, endo-therapeutic, surgical or radiological intervention to achieve hemostasis, re bleeding and mortality. Unfortunately, no single risk score has been shown to be accurate at measuring all relevant outcomes.

The most widely used score is Glasgow Blatchford "GBS" which is a pre endoscopic score. It is useful in prediction of therapeutic intervention for bleeding. More recently, other scores have been developed as ABC score which showed good performance for predicting mortality. MAP score highly predicted therapeutic intervention and mortality. H3B2 score predicted the need of urgent hemostasis.

Limited data are available on the validity of the new scoring systems in predicting the outcome of Egyptian non-cirrhotic patients with acute UGIB. Therefore, The investigators will conduct our study to shed some light on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Adult non cirrhotic patients
* patients more than 18 years old
* Hematemesis or coffee grounds vomiting.
* Melena with or without hematemesis.
* Blood in nasogastric tube in emergency unit.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients known to be cirrhotic.
* Patients presented with GIT bleeding but refuse to be examined by GIT endoscopy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients within the current study will be subjected to:
  I-Complete medical history. II-Through clinical examination. III-Laboratory investigations including Complete blood count (CBC) Liver profile (serum bilirubin, serum albumin, PT and INR) Blood urea and creatinine
  IV-Abdominal Ultrasonography :
  VI-Risk scoring systems :
  At the time of admission, each of following 4 scores will be calculated and recorded (Glasgow Blatchford score, MAP score, H3B2 score and ABC score to validate outcome in the studied patients The Glasgow-Blatchford score "GBS" (6) MAP score, (11) The ABC score: (10) H3B2 score (12)
  V-Upper GIT endoscopy :
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
correlation between Glasgow -Blatchford score, MAP score. | Baseline
  correlation between Glasgow -Blatchford score, MAP score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay.
correlation between Glasgow -Blatchford score, H3B2 score. | Baseline
  correlation between Glasgow -Blatchford score, H3B2 score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay.
correlation between Glasgow -Blatchford score, ABC score. | Baseline
  correlation between Glasgow -Blatchford score, ABC score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay.
correlation between MAP score, H3B2 score. | Baseline
  correlation between MAP score, H3B2 score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay .
correlation between MAP score, ABC score. | Baseline
  correlation between MAP score, ABC score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay.
correlation between H3B2 score, ABC score. | Baseline
  correlation between H3B2 score, ABC score regarding to Need of intervention, Re bleeding, Thirty-day mortality, length of hospital stay.

REFERENCES:
- [Background] Feinman M, Haut ER. Upper gastrointestinal bleeding. Surg Clin North Am. 2014 Feb;94(1):43-53. doi: 10.1016/j.suc.2013.10.004. PMID 24267496
- [Background] Elwakil R, Reda MA, Abdelhakam SM, Ghoraba DM, Ibrahim WA. Causes and outcome of upper gastrointestinal bleeding in Emergency Endoscopy Unit of Ain Shams University Hospital. J Egypt Soc Parasitol. 2011 Aug;41(2):455-67. PMID 21980783
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Blatchford O, Murray WR, Blatchford M. A risk score to predict need for treatment for upper-gastrointestinal haemorrhage. Lancet. 2000 Oct 14;356(9238):1318-21. doi: 10.1016/S0140-6736(00)02816-6. PMID 11073021
- [Background] Saltzman JR, Tabak YP, Hyett BH, Sun X, Travis AC, Johannes RS. A simple risk score accurately predicts in-hospital mortality, length of stay, and cost in acute upper GI bleeding. Gastrointest Endosc. 2011 Dec;74(6):1215-24. doi: 10.1016/j.gie.2011.06.024. Epub 2011 Sep 10. PMID 21907980
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Risk assessment after acute upper gastrointestinal haemorrhage. Gut. 1996 Mar;38(3):316-21. doi: 10.1136/gut.38.3.316. PMID 8675081
- [Background] Orpen-Palmer J, Stanley AJ. A Review of Risk Scores within Upper Gastrointestinal Bleeding. J Clin Med. 2023 May 26;12(11):3678. doi: 10.3390/jcm12113678. PMID 37297873
- [Background] Laursen SB, Oakland K, Laine L, Bieber V, Marmo R, Redondo-Cerezo E, Dalton HR, Ngu J, Schultz M, Soncini M, Gralnek I, Jairath V, Murray IA, Stanley AJ. ABC score: a new risk score that accurately predicts mortality in acute upper and lower gastrointestinal bleeding: an international multicentre study. Gut. 2021 Apr;70(4):707-716. doi: 10.1136/gutjnl-2019-320002. Epub 2020 Jul 28. PMID 32723845
- [Background] Redondo-Cerezo E, Vadillo-Calles F, Stanley AJ, Laursen S, Laine L, Dalton HR, Ngu JH, Schultz M, Jimenez-Rosales R. MAP(ASH): A new scoring system for the prediction of intervention and mortality in upper gastrointestinal bleeding. J Gastroenterol Hepatol. 2020 Jan;35(1):82-89. doi: 10.1111/jgh.14811. Epub 2019 Aug 19. PMID 31359521
- [Background] Sasaki Y, Abe T, Kawamura N, Keitoku T, Shibata I, Ohno S, Ono K, Makishima M. Prediction of the need for emergency endoscopic treatment for upper gastrointestinal bleeding and new score model: a retrospective study. BMC Gastroenterol. 2022 Jul 11;22(1):337. doi: 10.1186/s12876-022-02413-8. PMID 35820868